CLINICAL TRIAL: NCT01071473
Title: Resistance and Aerobic Exercise for Subclinical Anthracycline Cardiomyopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CARHAB
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Cardiomyopathy
Keywords: Childhood cancer; Anthracyclines; Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise Group (Other): Survivors of childhood cancer treated with anthracyclines and known to have cardiomyopathy will participate in a 12 week exercise intervention.
  Interventions: Other: 12 Week Exercise Intervention

INTERVENTIONS:
Other: 12 Week Exercise Intervention — Trial of a 12-week period of combined endurance and resistance training in survivors of childhood cancer who were treated with doxorubicin and/or daunorubicin and have impaired cardiac function.

SUMMARY:
This application proposes a prospective, single arm feasibility clinical trial of a 12-week period of combined endurance and resistance training in survivors of childhood cancer who were treated with doxorubicin and/or daunorubicin and have impaired cardiac function.

Baseline and post intervention imaging, laboratory, and neuropsychological evaluations will be used to determine the effects of the intervention on body composition, serum lipid profile, exercise tolerance, and neurocognitive functioning. Participants will be called weekly to monitor compliance with the intervention. Incentives will be given at intervals during the trial to optimize compliance with the intervention.

DETAILED DESCRIPTION:
This study will evaluate the feasibility of a 12-week exercise intervention on the cardiac function of survivors of childhood cancer treated with anthracyclines and known to have cardiomyopathy.

As a secondary objective, the study will document the effect of a 12-week exercise intervention on exercise tolerance, as determined by measurement of peak VO2 and peak exercise workload, shortening fraction, ejection fraction, and left ventricular wall thickness, and assess the impact of the intervention on neurocognitive functioning in survivors of childhood cancer treated with anthracyclines and known to have cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Treated at St. Jude Children's Research Hospital (SJCRH)
* Ages 0 - 17 years at time of treatment
* Treated for any type of cancer
* ≥ 10 years from date of diagnosis
* ≥ 2 years after completion of active cancer therapy
* ≥ 18 years of age
* Treated with doxorubicin and/or daunorubicin (any cumulative dose)
* Ejection fraction of < 55% without medications
* Does not currently meet the Centers for Disease Control (CDC) recommendations for exercise for adults

Exclusion Criteria:

* Ejection fraction ≤ 40%
* Pregnant females (Positive Urine pregnancy Test).
* History of congenital heart disease
* History of myocardial infarction
* History of acute coronary syndrome
* Individuals with pacemakers or implanted defibrillators
* History of radiation therapy that included any part of the heart
* ≥1-mm J-point depression (depression measured 80 msec after J-point) with ST segment flat or down-sloping in the majority of complexes in any ECG lead except AVR with exercise testing.
* All patients will be classified using the recommendations of the American Heart Association. Patients found to be in Class A, C or Class D will not be eligible for study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The primary aim of this proposal is to evaluate the feasibility of a 12-week exercise intervention among survivors of childhood cancer treated with anthracyclines and known to have cardiomyopathy. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Green, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org